CLINICAL TRIAL: NCT05440617
Title: Biorepository in Participants Who Undergo OTC for Gonadotoxic Therapy
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000715; 000715-CH
Record Dates: First submitted 2022-06-30; First posted 2022-07-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-08-29

CONDITIONS: Acute Ovarian Failure; Infertility; Early Menopause And Infertility In Females After Treatment For Childhood Cancer
Keywords: Ovarian Tissue Preservation; Cancer Survivors And Infertility; Acute Ovarian Failure In The Childhood Cancer Survivor Study; Ovarian Failure After Radiation; Natural History
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects Treated with Gonadotoxic therapy: Subjects who have planned to undergo OTC for gonadotoxic therapy based on current standard of care.

SUMMARY:
Background:

Medical advances have improved survival rates for many cancers and other illnesses. This means that more people are coping with the long-term effects of these treatments. Some treatments can cause female infertility. Ovarian tissue cryopreservation (OTC) may help. Before undergoing a treatment that may damage their fertility, patients may opt to freeze a sample of ovarian tissue. The tissue contains immature egg cells. When thawed, the tissue can be reimplanted. This procedure can help women become pregnant.

Objective:

This natural history study will create a databank of ovarian tissue. The NIH will provide OTC as a clinical service. The NIH will also request a portion of the tissue to use for research.

Eligibility:

Females aged 4 to 35 who opt to have OTC before receiving cancer treatment.

Design:

Participants will be screened. Their existing medical records will be reviewed.

They will be asked if they want to donate a portion of their ovarian tissue for research. No more than 20% of the tissue collected will be taken for research. Some other tissues that would otherwise be discarded will also be kept.

Medical data from each participant may also be collected and stored in the database. This data may include results of routine blood tests, imaging tests, and other information. The data will be coded for privacy.

Participants will answer a questionnaire. They will be asked about their fertility treatment and general health. The survey takes about 30 minutes.

They will repeat the questionnaire once a year for 30 years.

DETAILED DESCRIPTION:
Study Description:

We will provide ovarian tissue cryopreservation (OTC) as a clinical service at NIH and collect a portion of the tissue for research regarding normal histology and function of the human ovary. In addition, de-identified data will be entered in a national database which will allow future research regarding short term and long term complications (Including impact of therapy on remaining ovarian function), as well as long term outcomes including reproductive health outcomes (including rate of tissue reimplantation and pregnancies)

Objectives:

Primary objective: is to create a databank of human ovarian tissue to elucidate histology and function in human ovaries.

Secondary objective: will be to populate a national database of individuals who have undergone OTC in order to elucidate short and long term outcomes including complications and reproductive health parameters.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent/assent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Subjects who have planned to undergo OTC for gonadotoxic therapy based on current standard of care.

EXCLUSION CRITERIA:

-An individual who meets any of the following criteria will be excluded from participation in this study:

--Adults subjects with psychological, psychiatric, or other conditions which prevent giving fully informed consent.

Ages: 4 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects who will undergo gonadotoxic treatment at NCI.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2041-09-21 (Estimated); Study Completion 2041-09-21 (Estimated)

PRIMARY OUTCOMES:
create a databank of human ovarian tissue | end of study
  Create a databank of human ovarian tissue to elucidate histology and function in human ovaries

SECONDARY OUTCOMES:
create a databank of human ovarian tissue to elucidate histology and function in human ovaries | end of study
  Populate a national database of individuals who have undergone OTC in order to elucidate short and long term outcomes including complications and reproductive health parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Gomez-Lobo, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Patrizio P, Butts S, Caplan A. Ovarian tissue preservation and future fertility: emerging technologies and ethical considerations. J Natl Cancer Inst Monogr. 2005;(34):107-10. doi: 10.1093/jncimonographs/lgi023. PMID 15784838
- [Background] Sklar CA, Mertens AC, Mitby P, Whitton J, Stovall M, Kasper C, Mulder J, Green D, Nicholson HS, Yasui Y, Robison LL. Premature menopause in survivors of childhood cancer: a report from the childhood cancer survivor study. J Natl Cancer Inst. 2006 Jul 5;98(13):890-6. doi: 10.1093/jnci/djj243. PMID 16818852
- [Background] Chemaitilly W, Mertens AC, Mitby P, Whitton J, Stovall M, Yasui Y, Robison LL, Sklar CA. Acute ovarian failure in the childhood cancer survivor study. J Clin Endocrinol Metab. 2006 May;91(5):1723-8. doi: 10.1210/jc.2006-0020. Epub 2006 Feb 21. PMID 16492690
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000715-CH.html